CLINICAL TRIAL: NCT00152295
Title: A Phase II Long-Term Extension Safety Study of J867 Administered With Estrogen to Postmenopausal Women
Brief Title: A Long-Term Study to Evaluate the Safety of Asoprisnil and Estrogen Administration to Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M01-280
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Postmenopause
Keywords: Postmenopausal; Amenorrhea; Hormone replacement therapy; HRT; asoprisnil; Estrogen Replacement Therapy, postmenopause
MeSH Terms: conditions — Amenorrhea | interventions — asoprisnil; Estrogens, Conjugated (USP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil/Premarin

INTERVENTIONS:
Drug: Asoprisnil/Premarin — 10 mg (2-5mg tablets) asoprisnil and 0.625 mg Premarin tablets, oral daily for 6 months

SUMMARY:
The objective of this study is to determine the long-term safety of asoprisnil 10 mg when administered to postmenopausal women with Premarin® 0.625 mg

DETAILED DESCRIPTION:
The objective of this study is to determine the long-term safety of asoprisnil 10 mg (2-5mg tablets) when taken with Premarin® 0.625 mg, by postmenopausal women, for 6 months after an initial 12 weeks in Study M00-198. Pharmacodynamic effects to be assessed include uterine bleeding pattern, endometrial biopsy results, and endometrial thickness. Safety assessments will include clinical laboratory results, physical examination with vital signs, pelvic and breast examinations, ultrasound results, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of study M00-198
* Continued good general health
* Negative urine pregnancy test

Exclusion Criteria:

* History of known or suspected cancer other than basal cell carcinoma in last 5 years
* History of reproductive endocrine disorder
* Submucous or other symptomatic fibroid which would confound efficacy
* Ovarian mass
* Ongoing treatment with an excluded medication
* Stenosis of the cervix
* Any abnormal lab result the study-doctor considers significant.

Ages: 48 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2001-04; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
The percent of subjects in each endometrial biopsy diagnostic category summarized using SPRM Classification System. | Throughout Study
The percentage of subjects in each endometrial biopsy diagnostic category summarized using SPRM Classification System | Months 3,6
Change from baseline in endometrial thickness (mm) as measured by transvaginal ultrasound. | Months 3,6

SECONDARY OUTCOMES:
Frequency and amount of vaginal bleeding assessed via daily diary. | Throughout study
Frequency and severity of hot flushes assessed via daily diary. | Throughout study
Mean change from baseline in endocrine determinations. | Months 2,4,and 6
Global efficacy question | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott